CLINICAL TRIAL: NCT05373186
Title: A Trial Investigating the Pharmacodynamics of BC Combo THDB0207 Compared With Humalog® Mix25 and Simultaneous Injections of Humalog® and Lantus® in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CT046-ADO05
Record Dates: First submitted 2022-05-04; First posted 2022-05-13 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — Glucose Clamp Technique; Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Three-period crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BC Combo THDB0207 (Experimental): Single administration of BC Combo THDB0207
  Interventions: Drug: Euglycemic clamp with BC Combo THDB0207
- Humalog® Mix25 (Active Comparator): Single administration of Humalog® Mix25
  Interventions: Drug: Euglycemic clamp with Humalog® Mix25
- Humalog® and Lantus® (Active Comparator): Simultaneous administration of Humalog® and Lantus®
  Interventions: Drug: Euglycemic clamp with Humalog® and Lantus®

INTERVENTIONS:
Drug: Euglycemic clamp with BC Combo THDB0207 — Administration of a single dose of BC Combo THDB0207 during an euglycemic clamp procedure
  Arms: BC Combo THDB0207
Drug: Euglycemic clamp with Humalog® Mix25 — Administration of a single dose of Humalog® Mix25 during an euglycemic clamp procedure
  Arms: Humalog® Mix25
Drug: Euglycemic clamp with Humalog® and Lantus® — Simultaneous administration of Humalog® and Lantus® during an euglycemic clamp procedure
  Arms: Humalog® and Lantus®

SUMMARY:
This is a randomised, double-blind, double-dummy, active-controlled, three-period crossover euglycemic clamp trial in healthy Chinese volunteers.

Each subject will be randomly allocated to one of 6 treatment sequences. Each sequence comprises one single dose of BC Combo THDB0207, one single dose of Humalog® Mix25, or simultaneous administration of Humalog® and Lantus®.

Subjects will come in a fasted state to the clinical trial centre in the morning of each dosing day and stay at the clinical trial centre until the 30-hour clamp procedures have been terminated.

DETAILED DESCRIPTION:
Subjects will attend the study site in the morning in a fasted state and will be connected to an automated glucose clamp device (ClampArt). Prior to dose administration plasma glucose will be stabilised at a defined target level by means of an intravenous infusion of glucose or insulin. IMP administration will be done by an unblinded person by means of subcutaneous injections in the abdominal wall.

Following each dosing a euglycaemic glucose clamp procedure will be carried out for up to 30 hours.

The pharmacodynamic assessment will be based on the time course of glucose infusion rate (GIR) and plasma glucose.

Plasma insulin concentrations will be measured using a specific validated bioanalytical method differentiating concentrations of insulin glargine, of its main metabolites insulin-glargine-M1 and insulin-glargine M2, and of insulin lispro. Pharmacokinetic insulin assessments will be based on total insulin concentration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Chinese origin. To qualify as a subject of Chinese origin (first-generation Chinese), the subject, the subject's biological parents, and all of the subject's biological grandparents are of exclusive Chinese descent and have been born in China.
* BMI between 18.5 and 30.0 kg/m2, both inclusive.
* Fasting plasma glucose concentration <= 5.6 mmol/L (100 mg/dL).

Exclusion Criteria:

* Known or suspected hypersensitivity to IMP(s) or any of the excipients or to any component of the IMP formulation.
* Receipt of any investigational medicinal product within 3 months before randomisation in this trial.

Women of childbearing potential who are not using a highly effective contraceptive method.

* Any history or presence of a life-threatening disease (i.e. cancer except basal cell skin cancer or squamous cell skin cancer), or of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic (including type 1 and type 2 diabetes mellitus, haematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynaecologic (if female), or infectious disease, or signs of acute illness as judged by the investigator.
* Heart rate at rest outside the range of 50-90 beats per minute.
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
AUCGIR 0-2h | From t=0 to t=2 hours after IMP administration
  Area under the glucose infusion rate curve until 2 hours after IMP dosing

SECONDARY OUTCOMES:
AUCGIR 0-last | From t=0 to t= 30 hours after IMP administration
  Area under the glucose infusion rate curve from 0 hours until the end of clamp
GIRmax | From t=0 to t= 30 hours after IMP administration
  Maximum Glucose Infusion Rate
AUCGIR 0-1h | From t=0 to t=1 hours after IMP administration
  Area under the glucose infusion rate curve until 1 hour after IMP dosing
AUCGIR 0-6h | From t=0 to t=6 hours after IMP administration
  Area under the glucose infusion rate curve until 6 hours after IMP dosing
AUCGIR 0-24h | From t=0 to t=24 hours after IMP administration
  Area under the glucose infusion rate curve until 24 hours after IMP dosing
tGIRmax | From t=0 to t=30 hours after IMP administration
  Time to maximum glucose infusion rate
tonset of action | From t=0 to t=30 hours after IMP administration
  Time until plasma glucose (PG) has decreased by at least 5 mg/dL from the baseline PG value
AUCINSlast | From t=0 to t=30 hours after IMP administration
  Area under the insulin concentration-time curve from t=0 to the last measured insulin concentration above LLOQ
AUCINS 0-2h | From t=0 to t=2 hours after IMP administration
  Area under the insulin concentration-time curve during from t=0 to t=2h
AUCINS 0-6h | From t=0 to t=6 hours after IMP administration
  Area under the insulin concentration-time curve during from t=0 to t=6h
AUCINS 2-4h | From t=2 to t=4 hours after IMP administration
  Area under the insulin concentration-time curve during from t=2 to t=4h
AUCINS 6-12h | From t=6 to t=12 hours after IMP administration
  Area under the insulin concentration-time curve during from t=6 to t=12h
AUCINS 12-30h | From t=12 to t=30 hours after IMP administration
  Area under the insulin concentration-time curve during from t=12 to t=30h
AUCINS 0-30h | From t=0 to t=30 hours after IMP administration
  Area under the insulin concentration-time curve during from t=0 to t=30h
CmaxINS | From t=0 to t= 30 hours after IMP administration
  Maximum insulin concentration
Tonset ins | From t=0 to t=30 hours
  Tonset of insulin appearance
Adverse Events | From the first IMP administration to the follow-up visit (i.e. up to 11 weeks)
  Incidence of adverse events
Serious Adverse Events | From the first IMP administration to the follow-up visit (i.e. up to 11 weeks)
  Incidence of Serious Adverse Events
Local tolerability | From the first IMP administration to the follow-up visit (i.e. up to 11 weeks)
  Incidence of injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany